CLINICAL TRIAL: NCT01060540
Title: The Impact of Genetic Testing for Type 2 Diabetes on Health Behaviors
Brief Title: Genetic Testing for Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IBD 09-039
Record Dates: First submitted 2010-01-29; First posted 2010-02-02 (Estimated); Results first posted 2014-08-04 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Diabetes Mellitus
Keywords: genetic screening
MeSH Terms: conditions — Diabetes Mellitus | interventions — Genetic Testing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CR+G (Experimental): conventional risk counseling (lifetime risk, fasting plasma glucose, and family history) plus genetic testing for type 2 diabetes
  Interventions: Genetic: genetic testing for type 2 diabetes; Behavioral: Conventional risk counseling
- CR+EYE (Active Comparator): conventional risk counseling (lifetime risk, fasting plasma glucose, and family history) plus eye disease counseling
  Interventions: Behavioral: Conventional risk counseling; Behavioral: eye disease counseling

INTERVENTIONS:
Genetic: genetic testing for type 2 diabetes — TCF7L2, PPARG, or KCNJ11
  Arms: CR+G
Behavioral: Conventional risk counseling — Risk based on lifetime risk, fasting plasma glucose results, and family history.
Behavioral: eye disease counseling — addresses risk for age-related macular degeneration, glaucoma, cataracts
  Arms: CR+EYE

SUMMARY:
In this 6-month randomized, controlled trial, we examined whether providing participants with genetic test results and counseling regarding their risk for type 2 diabetes would motivate them to improve their health behaviors and lose weight to reduce their diabetes risk. We hypothesized that participants who received conventional diabetes counseling plus genetic test results and counseling would have at least 6 lb greater weight loss at 3 months than participants who received conventional diabetes counseling without genetic test results.

DETAILED DESCRIPTION:
In this 6-month randomized, controlled trial, we evaluated the impact of genetic testing for type 2 diabetes on psychological, health behavior, and clinical outcomes. Eligibility criteria included age 21 to 65 years, overweight or obese (body mass index [BMI] >27 kg/m2), and no prior diagnosis of type 2 diabetes. At baseline, participants (N=601) had conventional risk factors assessed, including demographics, fasting plasma glucose (FPG), and family history. They also provided blood samples for genetic testing of TCF7L2, PPARG, and KCNJ11, three genes that confer elevated risk for development of type 2 diabetes. Participants were then randomized to receive conventional counseling plus control eye disease counseling (CR+EYE) or conventional counseling plus genetic test results (CR+G). Two to four weeks following the baseline visit, when the genetic test results were available, participants returned for a visit with a genetic counselor. All participants received conventional risk counseling based on their lifetime population risk, FPG results, and family history. Next, participants were informed of their randomization assignments; CR+EYE participants received counseling on eye diseases, whereas CR+G participants received genetic counseling. Then perceived risk, affect, self-efficacy, and readiness to change were assessed. All other outcomes were also assessed at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* body mass index >27 kg/m2
* baseline fasting plasma glucose <=125 mg/dL

Exclusion Criteria:

* prior diagnosis of type 2 diabetes
* fasting plasma glucose >125 mg/dL on more than one occasion
* HbA1c > 7%
* taking diabetes medication
* actively losing weight
* enrolled in research study focusing on lifestyle changes
* unable to provide informed consent or answer survey questions unassisted
* residing in nursing home or receiving home health care
* active diagnosis of psychosis or dementia
* at least one error on 6-item cognitive screener

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 601 (Actual)
Dates: Start 2010-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corrine I. Voils, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

REFERENCES:
- [Result] Vorderstrasse AA, Cho A, Voils CI, Orlando LA, Ginsburg GS. Clinical utility of genetic risk testing in primary care: the example of Type 2 diabetes. Per Med. 2013 Aug;10(6):549-563. doi: 10.2217/pme.13.47. PMID 29776196
- [Result] Voils CI, Coffman CJ, Edelman D, Maciejewski ML, Grubber JM, Sadeghpour A, Cho A, McKenzie J, Blanpain F, Scheuner M, Sandelowski M, Gallagher MP, Ginsburg GS, Yancy WS Jr. Examining the impact of genetic testing for type 2 diabetes on health behaviors: study protocol for a randomized controlled trial. Trials. 2012 Aug 1;13:121. doi: 10.1186/1745-6215-13-121. PMID 22852560
- [Derived] Voils CI, Coffman CJ, Grubber JM, Edelman D, Sadeghpour A, Maciejewski ML, Bolton J, Cho A, Ginsburg GS, Yancy WS Jr. Does Type 2 Diabetes Genetic Testing and Counseling Reduce Modifiable Risk Factors? A Randomized Controlled Trial of Veterans. J Gen Intern Med. 2015 Nov;30(11):1591-8. doi: 10.1007/s11606-015-3315-5. Epub 2015 Apr 16. PMID 25876740
- [Derived] Waxler JL, O'Brien KE, Delahanty LM, Meigs JB, Florez JC, Park ER, Pober BR, Grant RW. Genetic counseling as a tool for type 2 diabetes prevention: a genetic counseling framework for common polygenetic disorders. J Genet Couns. 2012 Oct;21(5):684-91. doi: 10.1007/s10897-012-9486-x. PMID 22302620

RESULTS

PARTICIPANT FLOW:
Groups:
- CR+G: conventional risk counseling for type 2 diabetes (lifetime risk, fasting plasma glucose, and family history)
  results of genetic testing for type 2 diabetes based on the genes TCF7L2, PPARG, or KCNJ11
- CR+EYE: conventional risk counseling for type 2 diabetes (lifetime risk, fasting plasma glucose, and family history)
  eye disease counseling
Period: Overall Study
Arm/Group | CR+G | CR+EYE
Started | 303 | 298
Completed | 239 | 233
Not Completed | 64 | 65
Not completed — Withdrawal by Subject | 10 | 20
Not completed — Lost to Follow-up | 52 | 43
Not completed — Death | 2 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were calculated for all participants who attended the baseline session, where consent and baseline measures were obtained, regardless of whether they attended the intervention (risk counseling session).
Groups:
- Total: Total of all reporting groups
Arm/Group | CR+G | CR+EYE | Total
Number analyzed (Participants) | 303 | 298 | 601
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (9.1) | 54.4 (8.4) | 54.1 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 63 | 118
  Male | 248 | 235 | 483
Race/Ethnicity, Customized [Number; unit: participants]
  Non-Hispanic White | 137 | 115 | 252
  Other | 166 | 183 | 349
Region of Enrollment [Number; unit: participants]
  United States | 303 | 298 | 601
Education [Number; unit: participants]
  High school graduate or less | 82 | 72 | 154
  Some post-high school education | 221 | 226 | 447
Weight [Mean (Standard Deviation); unit: kg] | 103.8 (17.7) | 100.7 (18.9) | 101.8 (18.3)
Body mass index (BMI) stratification [Number; unit: participants]
  BMI >= 35 kg/m^2 | 95 | 85 | 180
  BMI<35 kg/m^2 | 208 | 213 | 421
Family history risk [Number; unit: participants]
  high | 79 | 60 | 139
  moderate | 79 | 94 | 173
  low | 141 | 140 | 281
  unknown | 4 | 4 | 8
Lifetime risk [Number; unit: participants]
  high | 213 | 193 | 406
  moderate | 81 | 99 | 180
  low | 8 | 5 | 13
  unknown | 1 | 1 | 2
Genetic risk [Number; unit: participants]
  high | 74 | NA — not tested | NA — Total not calculated because data are not available (NA) in one or more arms.
  moderate | 113 | NA — not tested | NA — Total not calculated because data are not available (NA) in one or more arms.
  low | 114 | NA — not tested | NA — Total not calculated because data are not available (NA) in one or more arms.
  unknown | 2 | NA — not tested | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Weight
Description: weight 3 months post-enrollment
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: kg
Groups:
- CR+G: conventional risk counseling (lifetime risk, fasting plasma glucose, and family history) plus genetic testing
  genetic testing for type 2 diabetes: TCF7L2, PPARG, or KCNJ11
- CR+EYE: conventional risk counseling (lifetime risk, fasting plasma glucose, and family history) plus control eye disease counseling
  Conventional risk counseling for type 2 diabetes: Conventional risk counseling: lifetime risk, fasting plasma glucose results, and family history.
Arm/Group | CR+G | CR+EYE
Number analyzed (Participants) | 303 | 298
kg | 103.8 (17.7) | 100.7 (18.9)
Statistical Analysis 1: Comparison: CR+G vs CR+EYE; Test type: Superiority or Other; p = 0.44, Mixed Models Analysis; Adjusted for family history (low/unknown vs. high/moderate) and BMI>=35 (yes vs no) stratification variables; Mean Difference (Net) = 0.2, 95% CI 2-sided [-0.3 to 0.7]

2. Secondary Outcome: Insulin Resistance (HOMA2-IR)
Description: Calculated using the updated homeostasis model assessment (HOMA) calculator at http://www.dtu.ox.ac.uk/homacalculator/
  Higher numbers indicate higher insulin resistance. There are no established cutoffs indicating impaired resistance.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CR+G | CR+EYE
Number analyzed (Participants) | 303 | 298
units on a scale | 4.1 (3.6) | 4.1 (4.5)
Statistical Analysis 1: Comparison: CR+G vs CR+EYE; Test type: Superiority or Other; p = 0.19, Mixed Models Analysis — adjusted for baseline BMI class and family history level stratification variables; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.1 to 0.3]

3. Secondary Outcome: Perceived Lifetime Risk of Type 2 Diabetes
Description: measured on 1-7 scale (definitely will not get diabetes to definitely will get diabetes)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CR+G | CR+EYE
Number analyzed (Participants) | 303 | 298
units on a scale | 3.1 (1.6) | 3.1 (1.6)
Statistical Analysis 1: Comparison: CR+G vs CR+EYE; Test type: Superiority or Other; p = 0.38, Mixed Models Analysis — adjusted for stratification variables baseline BMI and family history; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.4 to 0.1]

4. Secondary Outcome: Daily Caloric Intake
Description: Estimated daily caloric intake based on self-reported frequency and amount of intake of specific foods over the past 3 months as assessed by the Block Brief Food Frequency Questionnaire
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: kcal
Arm/Group | CR+G | CR+EYE
Number analyzed (Participants) | 303 | 298
kcal | 1487 (1127) | 1573 (894)
Statistical Analysis 1: Comparison: CR+G vs CR+EYE; Test type: Superiority or Other; p = 0.05, Mixed Models Analysis — adjusted for baseline family history and BMI; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.2 to 0.0]

5. Secondary Outcome: Moderate Intensity Physical Activity
Description: self-report based on the long version of the International Physical Activity Questionnaire. Moderate physical activity was queried in the domains of work (e.g., carrying light loads), transportation (e.g., bicycling), domestic chores and gardening (e.g., sweeping, raking), and leisure-time (e.g., bicycling, swimming).
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: minutes per week
Arm/Group | CR+G | CR+EYE
Number analyzed (Participants) | 303 | 298
minutes per week | 568 (650) | 633 (794)
Statistical Analysis 1: Comparison: CR+G vs CR+EYE; Test type: Superiority or Other; p = 0.68, generalized linear model for count data — adjusted for baseline family history and BMI; incident rate ratio = 0.9, 95% CI 2-sided [0.7 to 1.2]

ADVERSE EVENTS:
Arm/Group | CR+G | CR+EYE
Serious Adverse Events (participants affected / at risk) | 1/303 | 2/298
Other Adverse Events (participants affected / at risk) | 0/303 | 1/298
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CR+G (N=303) | CR+EYE (N=298)
Participant Death (General disorders) | 1 (1) | 1 (1) — Participant passed away as noticed in their electronic medical record as noted when trying to schedule a follow-up appointment. No cause was given.
Heart Attack (Cardiac disorders) | 0 (0) | 1 (1) — Participant had a heart attack and had a stent place. He was hospitalized for 4 days and sent home.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CR+G (N=303) | CR+EYE (N=298)
Syncope (General disorders) | 0 (0) | 1 (1) — Participant fainted during a blood draw at the lab.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes